CLINICAL TRIAL: NCT02629523
Title: A Phase II, Open-Label, Multicentre Study to Assess the Anti-tumour Activity of Afatinib in Patients With Activating Epidermal Growth Factor Receptor Mutation in Circulating Tumor DNA
Brief Title: Afatinib in Lung Cancer With EGFR Mutation From Circulating Tumor DNA
Acronym: LiquidLung-A
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chonnam National University Hospital (Other)
Responsible Party: Principal Investigator, Young-Chul Kim, Professor, Chonnam National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1200.271
Record Dates: First submitted 2015-12-10; First posted 2015-12-14 (Estimated); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Lung Neoplasms; EGFR Gene Mutation
MeSH Terms: conditions — Lung Neoplasms | interventions — Afatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Afatinib (Experimental): Treatment efficacy of afatinib will be assessed in patients with lung cancer harboring EGFR mutations which were detected from circulating tumor DNA.
  Interventions: Drug: Afatinib

INTERVENTIONS:
Drug: Afatinib — Treatment efficacy of afatinib will be assessed in patients with lung cancer harboring EGFR mutations which were detected from circulating tumor DNA.
  Other Names: Giotrif

SUMMARY:
Treatment efficacy of afatinib will be assessed in patients with lung cancer harboring EGFR mutations which were detected from circulating tumor DNA.

DETAILED DESCRIPTION:
Obtaining Tumor tissue or cytology samples are not always available in some patients with lung cancer. Recently, studies showed that circulating tumor DNA can be used as a suitable substitute for mutation analysis. The sensitivity of EGFR mutation tests using circulating tumor DNA was reported in the range of 65.7% (10) to 75% (11), with high specificity and positive predictive value. In this trial, treatment efficacy of afatinib will be assessed in patients with NSCLC harboring EGFR mutations which were detected from circulating tumor DNA.

ELIGIBILITY:
Inclusion Criteria:

1. Stage IIIB or IV lung cancer diagnosed radiologically with or without pathologic diagnosis
2. Age> 18 year-old
3. ECOG performance status 0~2.
4. Activating EGFR mutation (G719X, exon 19 deletion, L858R, L861Q) detected from circulating DNA
5. Any one of the following criteria should be met

   * Unavailable or failed pathologic/cytologic diagnosis
   * Wild type or failed EGFR testing based on tumor tissue
   * No more tumor sample available for EGFR test
6. Measurable lesion by RECIST v1.1
7. Females should be using adequate contraceptive measures, should not be breast feeding and must have a negative pregnancy test prior to start of dosing or evidence of non-child bearing potential.
8. Male patients should be willing to use barrier contraception.
9. Provision of signed and dated, written informed consent prior to any study specific procedures, sampling and analyses
10. Adequate organ function, defined as all of the following:

    * Absolute neutrophil count (ANC) >=1500/mm3
    * Platelet count >= 75,000 /mm3
    * Serum creatinine < 1.4 mg/dL
    * AST or ALT < three times the upper limit of normal

Exclusion Criteria:

1. Prior exposure to EGFR-TKI. Prior chemotherapy will be permitted.
2. Previous or concomitant malignancies at other sites, except effectively treated non-melanoma skin cancers, carcinoma in situ of the cervix, ductal carcinoma in situ or effectively treated malignancy that has been in remission for more than 3 years and is considered to be cured.
3. Severe or unstable medical conditions such as history or presence of clinically relevant cardiovascular abnormalities such as uncontrolled hypertension, congestive heart failure NYHA classification of ≥ 3, unstable angina or poorly controlled arrhythmia as determined by the investigator. Myocardial infarction within 6 months prior to randomisation.
4. Known pre-existing interstitial lung disease
5. Any history or presence of poorly controlled gastrointestinal disorders that could affect the absorption of the study drug (e.g. Crohn's disease, ulcerative colitis, chronic diarrhoea, malabsorption)
6. Active hepatitis B infection (defined as presence of HepB sAg and Hep B DNA), active hepatitis C infection (defined as presence of Hep C RNA) and/or known HIV carrier.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2020-05-11 (Actual)

PRIMARY OUTCOMES:
Efficacy evaluation RECIST v1.1 | 2 months
  Efficacy evaluation RECIST v1.1

SECONDARY OUTCOMES:
Progression Free Survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Young-Chul Kim, MD, PhD, Study Chair — Chonnam National University Hospital
Locations (1):
- Chonnam National University Hwasun Hospital, Hwasun, Jeollanam-do, South Korea

IPD SHARING:
Plan to Share IPD: No